CLINICAL TRIAL: NCT04783610
Title: Ethanol-induced Vestibular Dysfunction as a Model for Bilateral Vestibular Syndrome: Similarities in VHIT and VOG Data.
Brief Title: Ethanol-induced Vestibular Dysfunction as a Model for Bilateral Vestibular Syndrome.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Jussi Sarin, Clinical Teacher in the Department of Otorhinolaryngology, Turku University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202130409
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: vHIT- and VOG-model for Bilateral Vestibular Neuronitis
Keywords: vHIT; vestibular neuronitis; VOG
MeSH Terms: conditions — Vestibular Neuronitis | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study subjects for vHIT- and VOG-measurements (Experimental): Each study subject is his/hers own comparator at different phases of ethanol consumption.
  Interventions: Other: Ethanol

INTERVENTIONS:
Other: Ethanol — Ethanol will be administered via oral route.

SUMMARY:
The purpose of the study is to create a vHIT- and VOG-model for bilateral vestibular neuronitis, via ethanol administration in healthy human subjects.

DETAILED DESCRIPTION:
Ethanol administration has an effect on vestibular function, measurable with video head impulse test (vHIT)- and vestibulo-oculography (VOG)-methods.

The purpose of the study is to create a vHIT- and VOG-model for bilateral vestibular neuronitis, a disease with difficult diagnostics, via ethanol administration in healthy human subjects.

As subjects are consuming ethanol via oral route, vHIT-measurements and VOG-measurements (slow and rapid eye movement recordings) are being recorded in order to measure the change in vestibular function.

During approx. 5 hours, 4 vHIT measurements will take place, while subjects ingest ethanol towards 1 per mille levels, measured via alcoholmeter.

Necessary precautions include strict exclusion criteria regarding health of the subjects and also comprehensive preparedness for management of allergic reactions and other unusual phenomena related to alcohol consumption.

ELIGIBILITY:
Inclusion Criteria:

* no previous ear diseases
* normal hearing
* no signs of alcohol dependence (6 points or less in AUDIT-questionnaire)

Exclusion Criteria:

* previous ear diseases
* abnormal hearing
* signs of alcohol dependence (7 points or more in AUDIT-questionnaire)

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Ethanol-induced vestibular function decline as measured with vHIT-gain-value-measurements. | 5 hours or 1 work day
  Video head impulse test measures the speed of eye movement as well as head movement (degrees per second, taken from 60 ms time interval from the beginning of head movement), the latter being produced by the investigator. The ratio of a sudden horizontal head movement and a rapid eye movement towards the opposite direction (as the subject is trying to fixate gaze straight ahead) is referred as gain value. With succeeding measurements during ethanol consumption, gain values will be recorded. The data contains vHIT gain -values at base level, without ethanol consumption, as well as during and after ethanol consumption. The most important tool in statistical analysis of the data is repeated measures analysis of variance (rm ANOVA). This allows each test subject to act as his/hers own control, as succeeding measurements are being compared to the base line values. The statistical significance will be set at the p< 0.05 level.

IPD SHARING:
Plan to Share IPD: No